CLINICAL TRIAL: NCT06312124
Title: A Multi-Disciplinary Approach to the Opportunistic Salpingectomy for Primary Prevention of Ovarian Cancer
Brief Title: A Study of Opportunistic Salpingectomy to Prevent Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 24-006
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Surgery
Keywords: abdominal surgery; pelvic surgery; Opportunistic Salpingectomy; ovarian cancer prevention; 24-006; Memorial Sloan Kettering Cancer Center
MeSH Terms: interventions — Salpingectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants scheduled for non-gynecologic abdominopelvic surgery (Experimental): Participants will be aged ≥45 years, have at least 1 fallopian tube, will not desire or plan to have children in the future, and will be scheduled to undergo non-gynecologic abdominopelvic surgery.
  Interventions: Behavioral: Educational Module; Procedure: Salpingectomy

INTERVENTIONS:
Behavioral: Educational Module — Part 1 consists of an education module with premodule and postmodule assessment questionnaires.
Procedure: Salpingectomy — Part 2 consists of incorporating opportunistic salpingectomy /OS into non-gynecologic surgery

SUMMARY:
The purpose of this study is to find out how many participants are interested in a surgical preventive procedure after watching an educational video. Before and after watching the video, participants will complete questionnaires in the clinic.

ELIGIBILITY:
Inclusion Criteria:

Part I

* Age ≥45 years
* Scheduled visit with a nongynecologic surgeon
* Female or assigned female at birth

Part II

* Age ≥45 years
* At least one in situ fallopian tube
* No desire or plan to have children in the future
* Average risk of developing ovarian cancer

  ° Note: Average risk patients are defined as patients with no known genetic risk factor for developing ovarian cancer. Patients who, after obtaining family history, are suspected to have a hereditary ovarian cancer syndrome but have not yet been tested, will be referred for genetic evaluation.
* Planned nongynecologic, intraabdominal, or pelvic surgery
* Deemed to be a suitable candidate by gynecologic surgeon and primary nongynecologic surgeon (for example, on the basis of surgical history and current malignancy status)
* Approved and signed informed consent

Exclusion Criteria:

Part I

* Not fluent in English or Spanish

  ° If there is a non-english or non-spanish speaking participant who is a strong candidate and meets all other criteria for Part 2, they are able to go directly onto Part 2 without completing Part 1. (Please see additional details in section 4.1 and 7.0.)
* Known inherited ovarian cancer susceptibility

Part II

* Personal history of a gynecologic malignancy
* Carrier of a hereditary breast or ovarian cancer variant (e.g., BRCA1, BRCA2, BRIP1, PALB2, RAD51C, RAD51D, MLH1, MSH2, MSH6, PMS2)
* Suspicious ovarian, fallopian tube, or uterine lesion on preoperative imaging
* Previous bilateral salpingectomy or bilateral salpingo-oophorectomy
* Presence of ESSURE, or other tubal-implanted birth control at the time of surgery
* Current pregnancy
* Emergent procedure or emergency procedure that has to be completed within 24 hours where clinical consent occurs in the inpatient setting or where the patient's immediate well-being is in danger or condition may be life threatening
* Primary surgeon anticipates that OS will add significant time (>30-40min) to the planned procedure.
* Inability to access the pelvis (ex., patient prone/lateral position) during the planned procedure.
* Known history of pelvic fibrosis or significant adhesions.
* Procedures with palliative intent only

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2028-03-08 (Estimated); Study Completion 2028-03-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Opportunistic Salpingectomy/OS after completion of educational module | up to 2 years
  Evaluate the acceptance of Opportunistic Salpingectomy/OS among nongynecologic surgical patients after completion of an educational module

CONTACTS AND LOCATIONS:
Overall Officials: Kara Long Roche, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Johns Hopkins University (Data Collection Only), Baltimore, Maryland
  - Dana Farber Cancer Institute (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - MD Anderson Cancer Center (Data Collection Only), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org